CLINICAL TRIAL: NCT04957836
Title: Postoperative Respiratory Complications According to Neuromuscular Block Reversal With Sugammadex for Immediate Extubation in the Operating Room After Minimally Invasive Cardiac Surgery (MICS): a Retrospective Observational Study
Brief Title: Postoperative Respiratory Complications According to Neuromuscular Block Reversal After MICS
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2021-091
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Minimally Invasive Cardiac Surgery
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: reversal with sugammadex — reversal with sugammadex for immediate extubation in the operating room

SUMMARY:
Postoperative respiratory complications according to the type of drug (sugammadex, pyridostigmine) used for reversible neuromuscular block when extubating an endotracheal tube in the operating room after minimally invasive cardiac surgery, and the length of intensive care unit stay are going to be checked. Through these results, it will be investigated whether the use of rocuronium-sugarmadex for neuromuscular block and reversal in patients undergoing minimally invasive cardiac surgery is clinically useful.

DETAILED DESCRIPTION:
The enhanced recovery after surgery program (ERAS program) has been introduced across several surgical fields, and its benefits are well known, mainly in perioperative colorectal surgery, pancreatic surgery, urology and gynecology surgery. On the other hand, although there are suggestions for an early recovery program after surgery in the field of cardiac surgery, it is still in its infancy. Minimally invasive cardiac surgery has advantages over open thoracic surgery, such as faster recovery, less bleeding and transfusion, and a reduction in the frequency of arrhythmias, making it suitable for applying an early recovery program after surgery. For an early recovery program after surgery, a multidisciplinary approach is required throughout the surgery period, and among them, early endotracheal extubation, which has been emphasized before, is known to reduce hospital stay and mortality. In addition, such early endotracheal extubation includes extubation of the endotracheal tube in the operating room immediately after completion of surgery as well as within 6 hours of entering the intensive care unit after the end of surgery. For the reversibility of neuromuscular block, neostigmine, pyridostigmine, an acetylcholinesterase inhibitor, or sugammadex, a selective neuromuscular blocker binding agent, are mainly used. It is known to reduce the incidence of pulmonary complications. However, there is no study on the frequency of postoperative respiratory complications following neuromuscular block and reversibility using the Rocuronium-Sugarmadex combination in minimally invasive cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* In the case of an endotracheal tube extubation in the operating room among adult patients over the age of 18 who underwent minimally invasive cardiac surgery

Exclusion Criteria:

* Emergency surgery
* If the patient has severe uncontrolled lung disease
* In case of neuromuscular block using cisatracurium and rocuronium together
* When neuromuscular block and reversal using cysatracurium-pyridostigmine or rocuronium-sugammadex combinations are not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the case of an endotracheal tube extubation in the operating room among adult patients over the age of 18 who underwent minimally invasive cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Postoperative respiratory complications | from time point of extubation in the operating room to time point of transferring patient to general ward (up to 6 months)
  Postoperative respiratory complications

SECONDARY OUTCOMES:
the length of intensive care unit stay | during ICU hospitalization (up to 6 months)
  the length of intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea